CLINICAL TRIAL: NCT01013233
Title: Training of Cognitive Function of Patients After Chemotherapy
Brief Title: Cognitive Training to Improve Cognitive Function Following Chemotherapy
Acronym: KT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Freie Universität Berlin (Other)
Responsible Party: Fernando Dimeo, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KTST09
Record Dates: First submitted 2009-11-12; First posted 2009-11-13 (Estimated); Last update posted 2009-11-13 (Estimated); Status verified 2009-11

CONDITIONS: Cognitive Dysfunction
Keywords: cognitive dysfunction chemotherapy
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training; Sensitivity Training Groups; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- training (Experimental): Patients in this group start the cognitive training over 6 weeks directly after randomization.
  Interventions: Behavioral: cognitive training
- control (Placebo Comparator): In this control group begin the training in a cross-over design 7 weeks after randomization.
  Interventions: Other: control group

INTERVENTIONS:
Behavioral: cognitive training — cognitive training over 6 weeks, consist of 6 meetings (a 45minutes), three sessions focus on concentration tasks and three sessions on memory problems.
  Other Names: training group
  Arms: training
Other: control group — no intervention
  Other Names: controll group
  Arms: control

SUMMARY:
The purpose of this study is to improve cognitive dysfunction following chemotherapy, the investigators investigated to see whether a cognitive training for memory and concentration skills can improve cognitive performance in patients following cancer treatment.

DETAILED DESCRIPTION:
Patients following chemotherapy invited for a cognitive training. Before and after cognitive function will evaluate.

ELIGIBILITY:
Inclusion Criteria:

* patients with cancer 6 weeks after chemotherapy

Exclusion Criteria:

* patients with neurological or psychiatric disorders
* patients without compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
several cognitive tests (TAP, VLMT, TMT, Stroop, RWT, D2, LGT-3) | one weeks following the end of the cognitive training

SECONDARY OUTCOMES:
quality of life and subjective perception of cognitive problems | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Niedeggen, PhD, Principal Investigator — Freie Universität Berlin
Locations (1):
- Charite Universitätsmedizin Berlin, Berlin, State of Berlin, Germany